CLINICAL TRIAL: NCT05421741
Title: Prophylactic Antibiotic Coated Nail to Prevent Infection: A Clinical Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00086285; 01012022 (Other: Atrium Health); 40010222 (Other: Department of Defense)
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-06

CONDITIONS: Osteomyelitis Tibia; Tibial Fractures; Open Tibia Fracture
Keywords: Antibiotic-coated nail
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intramedullary Nail (Active Comparator): Traditional standard of care intramedullary (IM) nail
  Interventions: Other: Standard Intramedullary Nail
- Antibiotic Coated Intramedullary Nail (Active Comparator): Intramedullary Nail coated with 2 grams of vancomycin and 560 mg gentamicin liquid.
  Interventions: Drug: Antibiotic coated intramedullary Nail

INTERVENTIONS:
Drug: Antibiotic coated intramedullary Nail — Antibiotic coated intramedullary nail:
  A mixture of 40gm bag of acrylic cement, antibiotic powder (Vancomycin 2gm) and 560mg gentamicin liquid. The intramedullary is coated with the mixture using a cement gun tube.
  Other Names: Local Gentamicin 560 Powder; Vancomycin 2gm Liquid
  Arms: Antibiotic Coated Intramedullary Nail
Other: Standard Intramedullary Nail — Standard Intramedullary Nail
  Arms: Intramedullary Nail

SUMMARY:
This prospective randomized clinical trial will compare outcomes between patients treated primarily with a prophylactic antibiotic coated nail and those treated with traditional standard of care intramedullary (IM) nailing.

DETAILED DESCRIPTION:
Despite significant treatment advances and protocols to prevent infection, severe open fractures of the lower extremity still have very high rates of deep infection. Infection in an active duty military population increases disability and decreases the likelihood of returning to duty. In addition, infection is one of the main factors associated with rehospitalization. Further, deep infections have not only resulted in increased disability after injury, infection is implicated as one of the main factors in late amputation. Among service members, only 20-25% with a severe open tibia fracture are able to return to active duty. Novel techniques for reducing infection are needed. The proposed study addresses the focus area of fracture-related infections, specifically the prevention of infection.

This prospective randomized clinical trial will compare outcomes between patients treated primarily with a prophylactic antibiotic coated nail and those treated with traditional standard of care intramedullary (IM) nailing.

This prospective randomized clinical trial will compare outcomes between patients treated primarily with a prophylactic antibiotic coated nail and those treated with traditional standard of care intramedullary (IM) nailing.

The target population for the proposed study is patients with severe open tibia fractures (Type II or Type III) who require definitive fixation with intramedullary nail recruited from one of the participating sites during the index hospitalization.

One group will be treated prophylactically using an antibiotic coated intramedullary nail at time of definitive fixation (1CN), while the second group will be treated with traditional standard of care intramedullary nail without antibiotic-coating (SN).

Participant will be followed for 12 months (data capture including patient interviews and clinical data capture from the treatment team and medical record at baseline, 6 weeks, 3 months, 6 months, and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older
* Gustilo Type II or III open tibia fracture requiring definitive fixation with intramedullary nail

Exclusion Criteria:

* Less than 18 years of age
* Allergy to vancomycin or gentamicin
* Unable to speak English or Spanish
* Pregnant and lactating women
* Prisoner
* Unable to follow up for 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who develop deep surgical site infection (SSI) | Day 30 through month 12
  Number of participants in each group who develop SSI as defined by the criteria establish by the Centers for Disease Control and Prevention (CDC). The CDC criteria define deep as occurring within 30 or 90 days after the procedure. However, we will continue to follow patients for 12 months and document any infections and other complications during this period.

SECONDARY OUTCOMES:
Radiographic Union Scale in Tibial fractures (RUST) score | week 6, month 3, month 6, and month 12
  The RUST score ranges from a minimum score of 4 (definitely not healed) to a maximum score of 12 (completely healed). The final x-ray obtained within a 12-month period following injury will be uploaded to REDCap for review by a blinded panel of investigators from participating sites.
Percentage of Union | week 6, month 3, month 6 and month12
  Union is the gradual process of bone regeneration after a fracture. Percentage of Union, as determined by the treating surgeon, will be assessed via radiographs. Recorded by surgeon as yes/no answers.
Time to Union | week 6, month 3, month 6 and month12
  Captured in days
Average Time to Return to Work/Duty | week 6, month 3, month 6 and month12
  number of days
International Physical Activity Questionnaire (IPAQ) | week 6, month 3, month 6 and month12
  IPAQ measures the total amount of physical activity completed in a 7 day period by calculating the minutes per week in in each physical activity level domain (walking, moderate and vigorous) by a metabolic equivalent energy (MET) expenditure estimate.
  Walking = 3.3 x number of walking minutes x number of walking days Moderate activity= 4.0 x number activity minutes x number of days Vigorous activity = 8 x number of activity minutes x number of days Total = Walking MET-min/wk+moderate MET-min/wk+vigorous MET-min/wk
Number of Subjects Who Have Returned to Work | week 6, month 3, month 6 and month12
  Determined by asking whether subjects have returned to work
Number of Participants who Return to Operating Room (OR) | Month 12
PROMIS-29 Subscale--Physical Function | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means higher physical function.
PROMIS-29 Subscale--Physical Function: Anxiety | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of anxiety.
PROMIS-29 Subscale--Depression | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of depression.
PROMIS-29 Subscale--Fatigue | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of fatigue.
PROMIS-29 Subscale--Sleep Disturbance | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of sleep disturbance.
PROMIS-29 Subscale--Pain Interference | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher level of pain interference.
PROMIS-29 Subscale--Ability to Participate in Social Roles and Activities | week 6, month 3, month 6 and month12
  The PROMIS-29 scales will be scored using a T-score metric method. A score of 50 points represents the population average for each scale, and 10 points represent one standard deviation. Higher scores means a higher ability to participate in social roles and activities.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Hsu, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (14):
- United States (14):
  - University of Florida Gainesville, Gainesville, Florida
  - Florida Orthopaedic Institute, Temple Terrace, Florida
  - Atrium Health Navicent, Macon, Georgia
  - University of Kentucky, Lexington, Kentucky
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - Atrium Health Cabarrus, Concord, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Houston, Houston, Texas
  - San Antonio Military Medical Center, San Antonio, Texas
  - Carilion Clinic, Roanoke, Virginia
  - Valley Health System, Winchester, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Owens BD, Kragh JF Jr, Macaitis J, Svoboda SJ, Wenke JC. Characterization of extremity wounds in Operation Iraqi Freedom and Operation Enduring Freedom. J Orthop Trauma. 2007 Apr;21(4):254-7. doi: 10.1097/BOT.0b013e31802f78fb. PMID 17414553
- [Result] Burns TC, Stinner DJ, Mack AW, Potter BK, Beer R, Eckel TT, Possley DR, Beltran MJ, Hayda RA, Andersen RC, Keeling JJ, Frisch HM, Murray CK, Wenke JC, Ficke JR, Hsu JR; Skeletal Trauma Research Consortium. Microbiology and injury characteristics in severe open tibia fractures from combat. J Trauma Acute Care Surg. 2012 Apr;72(4):1062-7. doi: 10.1097/TA.0b013e318241f534. PMID 22491628
- [Result] Bosse MJ, MacKenzie EJ, Kellam JF, Burgess AR, Webb LX, Swiontkowski MF, Sanders RW, Jones AL, McAndrew MP, Patterson BM, McCarthy ML, Travison TG, Castillo RC. An analysis of outcomes of reconstruction or amputation after leg-threatening injuries. N Engl J Med. 2002 Dec 12;347(24):1924-31. doi: 10.1056/NEJMoa012604. PMID 12477942
- [Result] Napierala MA, Rivera JC, Burns TC, Murray CK, Wenke JC, Hsu JR; Skeletal Trauma Research Education Consortium (STReC). Infection reduces return-to-duty rates for soldiers with Type III open tibia fractures. J Trauma Acute Care Surg. 2014 Sep;77(3 Suppl 2):S194-7. doi: 10.1097/TA.0000000000000364. PMID 25159355
- [Result] Johnson EN, Burns TC, Hayda RA, Hospenthal DR, Murray CK. Infectious complications of open type III tibial fractures among combat casualties. Clin Infect Dis. 2007 Aug 15;45(4):409-15. doi: 10.1086/520029. Epub 2007 Jul 5. PMID 17638186
- [Result] Ficke JR, Pollak AN. Extremity War Injuries: Development of Clinical Treatment Principles. J Am Acad Orthop Surg. 2007 Oct;15(10):590-5. doi: 10.5435/00124635-200710000-00003. PMID 17916782
- [Result] Section 1: Preventing and Managing Infection and Other Complications After Orthopaedic Trauma. J Orthop Trauma. 2017 Apr;31 Suppl 1:S2. doi: 10.1097/BOT.0000000000000798. No abstract available. PMID 28323794
- [Result] Masini BD, Owens BD, Hsu JR, Wenke JC. Rehospitalization after combat injury. J Trauma. 2011 Jul;71(1 Suppl):S98-102. doi: 10.1097/TA.0b013e3182218fbc. PMID 21795886
- [Result] Huh J, Stinner DJ, Burns TC, Hsu JR; Late Amputation Study Team. Infectious complications and soft tissue injury contribute to late amputation after severe lower extremity trauma. J Trauma. 2011 Jul;71(1 Suppl):S47-51. doi: 10.1097/TA.0b013e318221181d. PMID 21795878
- [Result] Cross JD, Stinner DJ, Burns TC, Wenke JC, Hsu JR; Skeletal Trauma Research Consortium (STReC). Return to duty after type III open tibia fracture. J Orthop Trauma. 2012 Jan;26(1):43-7. doi: 10.1097/BOT.0b013e31821c0ec1. PMID 21885998
- [Result] Bratzler DW, Houck PM; Surgical Infection Prevention Guidelines Writers Workgroup; American Academy of Orthopaedic Surgeons; American Association of Critical Care Nurses; American Association of Nurse Anesthetists; American College of Surgeons; American College of Osteopathic Surgeons; American Geriatrics Society; American Society of Anesthesiologists; American Society of Colon and Rectal Surgeons; American Society of Health-System Pharmacists; American Society of PeriAnesthesia Nurses; Ascension Health; Association of periOperative Registered Nurses; Association for Professionals in Infection Control and Epidemiology; Infectious Diseases Society of America; Medical Letter; Premier; Society for Healthcare Epidemiology of America; Society of Thoracic Surgeons; Surgical Infection Society. Antimicrobial prophylaxis for surgery: an advisory statement from the National Surgical Infection Prevention Project. Clin Infect Dis. 2004 Jun 15;38(12):1706-15. doi: 10.1086/421095. Epub 2004 May 26. PMID 15227616
- [Result] Pinto D, Manjunatha K, Savur AD, Ahmed NR, Mallya S, Ramya V. Comparative study of the efficacy of gentamicin-coated intramedullary interlocking nail versus regular intramedullary interlocking nail in Gustilo type I and II open tibia fractures. Chin J Traumatol. 2019 Oct;22(5):270-273. doi: 10.1016/j.cjtee.2019.03.006. Epub 2019 Jun 21. PMID 31443939
- [Result] Schmidmaier G, Kerstan M, Schwabe P, Sudkamp N, Raschke M. Clinical experiences in the use of a gentamicin-coated titanium nail in tibia fractures. Injury. 2017 Oct;48(10):2235-2241. doi: 10.1016/j.injury.2017.07.008. Epub 2017 Jul 10. PMID 28734495
- [Result] Jorge-Mora A, Amhaz-Escanlar S, Fernandez-Pose S, Garcia-Iglesias A, Mandia-Mancebo F, Franco-Trepat E, Guillan-Fresco M, Pino-Minguez J. Commercially available antibiotic-laden PMMA-covered locking nails for the treatment of fracture-related infections - A retrospective case analysis of 10 cases. J Bone Jt Infect. 2019 Jul 5;4(4):155-162. doi: 10.7150/jbji.34072. eCollection 2019. PMID 31555500
- [Result] Shiels SM, Mangum LH, Wenke JC. Revisiting the "race for the surface" in a pre-clinical model of implant infection. Eur Cell Mater. 2020 Jan 29;39:77-95. doi: 10.22203/eCM.v039a05. PMID 31995226
- [Result] Lin WT, Tan HL, Duan ZL, Yue B, Ma R, He G, Tang TT. Inhibited bacterial biofilm formation and improved osteogenic activity on gentamicin-loaded titania nanotubes with various diameters. Int J Nanomedicine. 2014 Mar 7;9:1215-30. doi: 10.2147/IJN.S57875. eCollection 2014. PMID 24634583
- [Result] Mauffrey C, Butler N, Hake ME. Fabrication of an Interlocked Antibiotic/Cement-Coated Carbon Fiber Nail for the Treatment of Long Bone Osteomyelitis. J Orthop Trauma. 2016 Aug;30 Suppl 2:S23-4. doi: 10.1097/BOT.0000000000000587. PMID 27441930
- [Result] Thonse R, Conway J. Antibiotic cement-coated interlocking nail for the treatment of infected nonunions and segmental bone defects. J Orthop Trauma. 2007 Apr;21(4):258-68. doi: 10.1097/BOT.0b013e31803ea9e6. PMID 17414554
- [Result] Barger J, Fragomen AT, Rozbruch SR. Antibiotic-Coated Interlocking Intramedullary Nail for the Treatment of Long-Bone Osteomyelitis. JBJS Rev. 2017 Jul;5(7):e5. doi: 10.2106/JBJS.RVW.16.00095. No abstract available. PMID 28719401
- [Result] O'Toole R, Joshi M, Carlini A, et al. Multicenter Randomized Trial Evaluating Intrawound Vancomycin Powder for Reducing Surgical Site Infection After Fracture Surgery. Orthopaedic Trauma Association; 2018; Orlando, FL
- [Result] Caroom C, Tullar JM, Benton EG Jr, Jones JR, Chaput CD. Intrawound vancomycin powder reduces surgical site infections in posterior cervical fusion. Spine (Phila Pa 1976). 2013 Jun 15;38(14):1183-7. doi: 10.1097/BRS.0b013e31828fcfb5. PMID 23474597
- [Result] Carver DC, Kuehn SB, Weinlein JC. Role of Systemic and Local Antibiotics in the Treatment of Open Fractures. Orthop Clin North Am. 2017 Apr;48(2):137-153. doi: 10.1016/j.ocl.2016.12.005. Epub 2017 Jan 30. PMID 28336038
- [Result] O'Toole RV, Joshi M, Carlini AR, Murray CK, Allen LE, Scharfstein DO, Gary JL, Bosse MJ, Castillo RC; METRC. Local Antibiotic Therapy to Reduce Infection After Operative Treatment of Fractures at High Risk of Infection: A Multicenter, Randomized, Controlled Trial (VANCO Study). J Orthop Trauma. 2017 Apr;31 Suppl 1:S18-S24. doi: 10.1097/BOT.0000000000000801. PMID 28323797
- [Result] Hanssen AD, Osmon DR, Patel R. Local antibiotic delivery systems: where are we and where are we going? Clin Orthop Relat Res. 2005 Aug;(437):111-4. No abstract available. PMID 16056035
- [Result] Shiels SM, Tennent DJ, Lofgren AL, Wenke JC. Topical rifampin powder for orthopaedic trauma part II: Topical rifampin allows for spontaneous bone healing in sterile and contaminated wounds. J Orthop Res. 2018 Dec;36(12):3142-3150. doi: 10.1002/jor.24155. Epub 2018 Oct 29. PMID 30270538
- [Result] Tennent DJ, Shiels SM, Sanchez CJ Jr, Niece KL, Akers KS, Stinner DJ, Wenke JC. Time-Dependent Effectiveness of Locally Applied Vancomycin Powder in a Contaminated Traumatic Orthopaedic Wound Model. J Orthop Trauma. 2016 Oct;30(10):531-7. doi: 10.1097/BOT.0000000000000617. PMID 27124826
- [Result] Shiels SM, Tennent DJ, Wenke JC. Topical rifampin powder for orthopedic trauma part I: Rifampin powder reduces recalcitrant infection in a delayed treatment musculoskeletal trauma model. J Orthop Res. 2018 Dec;36(12):3136-3141. doi: 10.1002/jor.24055. Epub 2018 Oct 5. PMID 29781552
- [Result] Berger ML, Dreyer N, Anderson F, Towse A, Sedrakyan A, Normand SL. Prospective observational studies to assess comparative effectiveness: the ISPOR good research practices task force report. Value Health. 2012 Mar-Apr;15(2):217-30. doi: 10.1016/j.jval.2011.12.010. PMID 22433752
- [Result] Dreyer NA, Tunis SR, Berger M, Ollendorf D, Mattox P, Gliklich R. Why observational studies should be among the tools used in comparative effectiveness research. Health Aff (Millwood). 2010 Oct;29(10):1818-25. doi: 10.1377/hlthaff.2010.0666. PMID 20921481
- [Result] Centers for Disease Control and Prevention. Surgical Site Infection (SSI) Event, January 2018. National Healthcare Safety Network. 2018
- [Result] Berrios-Torres SI, Umscheid CA, Bratzler DW, Leas B, Stone EC, Kelz RR, Reinke CE, Morgan S, Solomkin JS, Mazuski JE, Dellinger EP, Itani KMF, Berbari EF, Segreti J, Parvizi J, Blanchard J, Allen G, Kluytmans JAJW, Donlan R, Schecter WP; Healthcare Infection Control Practices Advisory Committee. Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection, 2017. JAMA Surg. 2017 Aug 1;152(8):784-791. doi: 10.1001/jamasurg.2017.0904. PMID 28467526
- [Result] Whelan DB, Bhandari M, Stephen D, Kreder H, McKee MD, Zdero R, Schemitsch EH. Development of the radiographic union score for tibial fractures for the assessment of tibial fracture healing after intramedullary fixation. J Trauma. 2010 Mar;68(3):629-32. doi: 10.1097/TA.0b013e3181a7c16d. PMID 19996801
- [Result] Kooistra BW, Dijkman BG, Busse JW, Sprague S, Schemitsch EH, Bhandari M. The radiographic union scale in tibial fractures: reliability and validity. J Orthop Trauma. 2010 Mar;24 Suppl 1:S81-6. doi: 10.1097/BOT.0b013e3181ca3fd1. PMID 20182243
- [Result] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Result] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Result] Cella D, Yount S, Rothrock N, Gershon R, Cook K, Reeve B, Ader D, Fries JF, Bruce B, Rose M; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS): progress of an NIH Roadmap cooperative group during its first two years. Med Care. 2007 May;45(5 Suppl 1):S3-S11. doi: 10.1097/01.mlr.0000258615.42478.55. PMID 17443116
- [Result] Schalet BD, Rothrock NE, Hays RD, Kazis LE, Cook KF, Rutsohn JP, Cella D. Linking Physical and Mental Health Summary Scores from the Veterans RAND 12-Item Health Survey (VR-12) to the PROMIS((R)) Global Health Scale. J Gen Intern Med. 2015 Oct;30(10):1524-30. doi: 10.1007/s11606-015-3453-9. Epub 2015 Jul 16. PMID 26179820
- [Result] Selim AJ, Rogers W, Fleishman JA, Qian SX, Fincke BG, Rothendler JA, Kazis LE. Updated U.S. population standard for the Veterans RAND 12-item Health Survey (VR-12). Qual Life Res. 2009 Feb;18(1):43-52. doi: 10.1007/s11136-008-9418-2. Epub 2008 Dec 3. PMID 19051059